# Supplementary Oxygen in Surgical and Medical wards evaluated by 30-day Mortality (SOSAM)

FULL STUDY PROTOCOL AND STATISTICAL ANALYSIS PLAN

# **INTRODUCTION**

### **OBJECTIVE**

The aim of this study is to investigate oxygen treatment and its correlation with morbidity and mortality in hospitalized medical and post-operative patients, the primary outcome being 30-day mortality.

Hyperoxia is hypothesized to increase 30-day mortality due to previous research indicating elevated arterial oxygenation as a negative predictor for mortality outcomes in various patient groups.

# **BACKGROUND**

Supplementary oxygen is widely used to both treat and prevent hypoxia in a clinical hospital setting. In spite of the widespread use of oxygen, and the well-known malicious effects of hypoxia, little is known about the harmful effects of abundant oxygen supply during hospital admission. Several methods of action have been proposed for the mechanism of harmful effects of hyperoxia, and studies have found hyperoxia to be harmful on a cellular level 1,2

Studies conducted on selected groups of patients have shown a harmful effect of short-term exposure of hyperoxia. Patients undergoing abdominal operations have been shown to have an increased long term-mortality when exposed to high levels of perioperative inspiratory oxygen<sup>3,4</sup> and patients with ST-elevation-myocardial infarction appear to have an increase in their level of myocardial injury after being randomized to high levels of supplementary oxygen.<sup>5</sup> It has been pointed out, that further research into this topic is of high relevance, seeing the current randomized controlled trials have focused mainly on the benefits of oxygen, rather than the potiential harmful effects of hyperoxia.<sup>6,7</sup>

# **METHODS**

### STUDY DESIGN

This study is designed as an observational retrospective cohort study, using a database consisting of data from the National Early Warning Score (EWS) from approximately 170.000 patients during hospitalization in the Capital Region of Denmark.

### SETTING

Regular measurements of NEWS-values on patients admitted to a hospital in the Capital region of Denmark has been standard practice since 2013. Data from NEWS-recordings on patients admitted to hospital in the period from 1 January 2014 to 31 December 2014 in the Capital Region of Denmark have previously been critically assessed and sanitized for unreliable entries. These sanitized recordings, combined with the primary diagnosis and 30-day mortality linked by the Danish CPR-number, are the primary datasets in this study.

Secondary analyses will be carried out on existing data for blood samples collected during hospital admission, and data for readmissions, ICU-admissions and reoperations.

### **PARTICIPANTS**

### **INCLUDED PATIENTS**

Patients are included according to the following criteria:

- Admission date (medical patients) or end of operation date (surgical patients) between 1<sup>st</sup> of January 2014 to 29<sup>th</sup> of December 2014.
- Age: ≥18
- Unique (first) admission for either:

### **Surgical Patients:**

Admitted for:

- Major operation with significant perforation of the peritoneum (laparotomy)
- Admission diagnosis (primary diagnosis) of hip fracture (DS720-DS722) combined with a surgical procedure code starting with KNF (hip surgery) for the same admission.

| DS720 | Fracture of neck of femur |
|-------|---------------------------|
| DS721 | Pertrochanteric fracture |
| DS722 | Subtrochanteric fracture |

# **Medical patients:**

Admitted under the primary diagnosis of:

• COPD with either acute exacerbation (DJ441) or acute lower respiratory infection (DJ440)

| DJ440 | Chronic obstructive pulmonary disease with acute lower respiratory infection |
|---|---|
| DJ441 | Chronic obstructive pulmonary disease with acute exacerbation, unspecified |

• Acute myocardial infarction (DI21X)

| DI21 | Acute myocardial infarction |
|--------|------------------------------------------------------------------|
| DI210 | Acute transmural myocardial infarction of anterior wall |
| DI210A | Anterior non-ST-elevation acute transmural myocardial infarction |
| DI210B | Anterior ST-elevation acute transmural myocardial infarction |
| DI211 | Acute transmural myocardial infarction of inferior wall |
| DI211A | Inferior non-ST-elevation Acute transmural myocardial infarction |
| DI211B | Inferior ST-elevation Acute transmural myocardial infarction |
| DI212 | Acute transmural myocardial infarction of other sites |
| DI213 | Acute transmural myocardial infarction of unspecified site |
| DI214 | Acute subendocardial myocardial infarction |
| DI219 | Acute myocardial infarction, unspecified |

### **EXCLUDED PATIENTS**

Patients are excluded according to the following criteria:

- No data on saturation within 48 hours after
  - Admission (Medical patients)
  - Discharge from the post anaesthesia care unit, PACU (Surgical patients)
- No data on primary outcome (30-day mortality)

A patient inclusion diagram will be included in the final manuscript. See below figure for proposed illustration.

### PATIENT INCLUSION DIAGRAM



Figure 1 - Overview of patient inclusion

### **VARIABLES**

As the majority of patients do not have a regular measurement of  $PaO_2$ , the exposure to hyperoxia will be estimated by combining the  $O_2$ -saturation (SpO2) as measured by pulse oximetry

and the amount of oxygen administration (measured in litres/min), both values obtained during the recording of EWS values.

Patients will be classified into three groups based on their oxygenation level. Patients will be assigned to the group according to which they spend the majority of time during the first 48 hours after either hospital admission for medical patients *or* discharge from the post anaesthesia care unit (PACU) for surgical patients. Patients previously diagnosed with COPD have a different setpoint for blood oxygenation, these patients are therefore classified according to the international guidelines for oxygenation in COPD-patients. Table 1 depicts the detailed classification of the three groups.

| | Нурохіа | Normoxia | Hyperoxia |
|---|---|---|---|
| Non-COPD | SpO2 <94% irrespective of | SpO2 94-98% in combination with | SpO2 >98% in combination with |
| | supplemental oxygen | supplemental oxygen | supplemental oxygen |
| | | <u>Or</u> | |
| | | SpO2 ≥94% without supplemental oxygen. | |
| COPD | SpO2 <88% irrespective of | SpO2 88-92% in combination with | SpO2 >92% in combination with |
| | supplemental oxygen | supplemental oxygen | supplemental oxygen |
| | | <u>Or</u> | |
| | | SpO2 ≥88% without supplemental oxygen. | |

Table 1 – Classification of oxygenation

Due to EWS measurements not being a function of time, a calculation will be done in order to estimate the weight of the individual EWS-measurement.

Based on the frequency of the EWS-measurements one measurement will be given a value corresponding to the fraction of time in the 48-hour period it covers, thus making it possible to estimate the oxemia status for the entire 48-hour period.

The normoxia group will serve as reference group for the analysis of the following outcome parameters in order to evaluate the effects of hyperoxia (primary analysis) and hypoxia (supplemental analysis):

The primary outcome is 30-day mortality, with secondary analysis of length of hospital stay, as well as the 30-day occurrence of admission to the Intensive Care Unit, re-operations and hospital readmission.

We will also assess associations of hyperoxia to organ-markers of disease severity: CRP (inflammation), creatinine (acute kidney injury) and troponin (myocardial injury), which will be

analysed by the peak level of each organ marker within 30 days.

As a supplemental analysis, we will also assess the clinical effects among patients with at least one arterial blood gas analysis during the 48 hours observation window, in which we divide patients in groups of hypoxia (PaO2 <8 kPa), normoxia (PaO2 8-12 kPa) and hyperoxia (PaO2 ≥12 kPa), according to the highest measured PaO2. We will also do a sensitivity analysis reassessing the

effect when patients are reassigned to groups according to exposure to hypoxia ≥8 hours or

hyperoxia ≥8 hours.

**DATA SOURCES** 

This study will be based on data from a National Early Warning Score (EWS) database recorded on

all patients hospitalized from 1 January 2014 to 31 December 2014 in the Capital Region. Data

Protection approval and Ethics Committee waiver have been approved for these data. The data

has been thoroughly validated for accurate entries and consists of data from approximately

170.000 unique hospital admissions in the Capital Region of Denmark.<sup>8</sup> Furthermore, the unique

CPR registration of all Danish patients, enables the analysis of organ markers within 30-days as

well as arterial blood gas in the previously defined 48-hour period.

**BIASES** 

The measurements of patients EWS-scores have all been manually registered and entered in the

EWS-database. Previous analyses of the EWS Database show inaccuracies in the entries with a bias

towards "normalized" values of vital parameters. Furthermore, EWS-measuring in the capital

region of Denmark was optional on patients at an "end of life pathway", potentially distorting the

data by not including the most critically ill patients.

The classification of patients according to their state of oxygenation was based on SpO2 measured

on a plethysmograph. Although such measurements correlate with the actual saturation of the

blood, factors such as peripheral circulation and nutritional status can effect this measurement

and thus affect the initial data.

POWER CALCULATION

MORTALITY

Hannibal Troensegaard 25/07-2018

The 30 day mortality in each of the four patient groups is estimated in order to calculate the power of the proposed study:

# A - Acute myocardial infarction: A = 7.5

Note: Estimated from a Prospective analysis on Danish patients with AMI. <sup>9</sup>

### **B** - **COPD** with exacerbation: B = 10%

Note: Estimated from a Danish study on COPD patients admitted with exacerbation with or without pneumonia (8,3-12,1%). <sup>10</sup>

# **C** - Hip fracture and surgery: C = 10%

Note: Estimated from a nationwide, population-based cohort study using prospectively collected data from the Danish Multidisciplinary Hip Fracture Registry, reporting 7,3 – 10% 30- day mortality on all admissions for hip fracture. Due to selection of patients WITH surgery in the proposed study, the 30-day mortality is expected to be towards the higher end, maybe higher, than the range referenced in the study. <sup>11</sup>

# **D** – Major abdominal surgery: D = 3.5%

Note: 30- day mortality estimated from the 30-day mortality in the PROXI-trial (2,9-4,4%). 12

### WEIGHTED AVERAGE OF 30-DAY MORTALITY:

Preliminary analysis suggests the following population sizes:

| | А | В | С | D | TOTAL |
|---|---|---|---|---|---|
| Pop size $(N_x)$ | $N_A = 2300$ | $N_B = 3100$ | $N_C = 2100$ | $N_D = 4600$ | 12100 |
| Mortality $(P_x)$ | $P_A = 7,5\%$ | $P_B = 10\%$ | $P_C = 10\%$ | $P_D = 3.5\%$ | |

Weighted average 30-day mortality:

$$\bar{P} = \frac{P_A * N_A + P_B * N_B + P_C * N_C + P_D * N_D}{N_A + N_B + N_C + N_D} \approx 7\%$$

POWER ON BASIS OF PRESUMED CLINICAL EFFICACY OF OXYGEN-GROUP

Values according to Figure 15.2, page 456 in "Practical Statistics for Medical Research" See appendix 1.

| Presumed difference in 30-day mortality between | Standardized difference | Power at N=10.000 patients |
|---|---|---|
| hyperoxia and normoxia | $P_1 - P_2$ | (derived from Figure 15.2, |
| (if N1-N2=0) | $\overline{\sqrt{ar{P}(1-ar{P})}}$ | Appendix 1) |
| $P_1 - P_2 = P$ | | |
| 7,25% - 6,75% = 0,5% | 0,0196 | 0,17 |
| 7,50% - 6,50% = 1,0% | 0,0392 | 0,42 |
| 7,75% - 6,25% = 1,5% | 0,0588 | 0,80 |
| 8,00% - 6,00% = 2,0% | 0,0784 | 0,97 |
| 8,25% - 5,75% = 2,5% | 0,0980 | >0,995 |
| 8,50% - 5,50% = 3,0% | 0,1176 | >0,995 |

### **WEAKNESSES OF THIS POWER CALCULATION**

The only patient population corresponding geographically to the currently proposed sample is the group from the PROXI trial used in group "D – major abdominal surgery". The other three mortality rates are from comparable but not exact same population base.

The power of the study was derived from a nomogram (Appendix 1) and not calculated with a formula, thus leaving room for reading errors.

Furthermore, the power calculation assumes the patient count in normoxia and hyperoxia are equal.

### **CONCLUSION**

With 12000 patients included in this study we have 80% power to detect a statistically significant difference in 30-day mortality of absolute risk reduction of 1.5% (relative risk reduction 19%) assuming the average 30-day mortality of the study sample is 7%, a distribution of patients 1:1 in the two groups and a significance level of 5%.

# PLAN FOR STATISTICAL ANALYSIS

### SUGGESTED DESCRIPTIVE DATA

Descriptive data for the population will be presented in table 1. For each of the three exposure groups, the following will be reported to characterise the study population: Age (mean), sex (percentage female), admission-hospital distribution and patient inclusion group distribution. The average EWS value (adjusted for chronic values) will also be included in the population description table.

| | | Нурохіа | Normoxia | Hyperoxia |
|-------------------|----------|---------|----------|-----------|
| Age (yr) | | | | |
| Sex (F%) | | | | |
| Hospital | | | | |
| | RH (%) | | | |
| | BFH (%) | | | |
| | GLO (%) | | | |
| | XX (%) | | | |
| Patient G | roup | | | |
| | MI (%) | | | |
| | COPD (%) | | | |
| | HIP (%) | | | |
| | ABD (%) | | | |
| Average EWS Value | | | | |

### **O**UTCOME DATA

Outcome data will be presented in table 2. The table will contain the three exposure groups and outcome data as calculated for each of the groups.

The primary outcome, 30 day mortality, is a binary variable for the individual patient, and will be reported as a fraction of positives within the exposure group population.

Length of stay and highest values for organ markers during the 30-day period will be treated as continuous variables with a non-normal distribution, and thus the median, not the mean, will be reported for these outcomes.

30-day admission to ICU, 30-day reoperation and 30-day readmission will be reported as a fraction of positives within the exposure group population.

Hannibal Troensegaard 25/07-2018

| GROUP | Mortality 30 d | Length of stay | Adm. ICU 30 d | Reop. 30 d | Readm. 30 d | Blood 30 d |
|---|---|---|---|---|---|---|
| Нурохіа | | | | | | CRP |
| | | | | | | Creatinine |
| | | | | | | Troponine |
| Normoxia | | | | | | CRP |
| | | | | | | Creatinine |
| | | | | | | Troponine |
| Hyperoxia | | | | | | CRP |
| | | | | | | Creatinine |
| | | | | | | Troponine |

For patients with least one arterial blood gas analysis during the 48 hours observation window, a secondary table will be reported, in which patients are divided in groups of hypoxia (PaO2 <8 kPa), normoxia (PaO2 8-12 kPa) and hyperoxia (PaO2 ≥12 kPa), according to their highest measured PaO2.

| GROUP | Mortality 30 d | Length of | Adm. ICU 30 | Reop. | Readm. | Blood 30 d |
|---|---|---|---|---|---|---|
| | | stay | | 30 d | 30 d | |
| Hypoxia PaO2 <8 kPa | | | | | | CRP |
| | | | | | | Creatinine |
| | | | | | | Troponine |
| Normoxia PaO2 8-12 kPa | | | | | | CRP |
| | | | | | | Creatinine |
| | | | | | | Troponine |
| Hyperoxia PaO2 ≥12 kPa | | | | | | CRP |
| | | | | | | Creatinine |
| | | | | | | Troponine |

### ANALYSES:

All outcome data will be compared in the normoxia vs. hyperoxia groups data and reported as an odds ratio in the primary analysis. 95% confidence intervals and the p-value will be reported for each outcome parameter. All values, including non-significant values, will be included in the final reporting.

Normoxia Hyperoxia Odds Ratio P value (95% CI)

Primary Outcome
30 day mortality

Secondary outcomes:
Adm. ICU 30 d
Reop. 30 d
Readm. 30 d
Blood 30 d
CRP
Creatinine
Troponine

# **O**THER ANALYSES

Secondary analyses will be carried out on normoxia vs hypoxia patients with the same outcome parameters as the primary analysis.

| | Нурохіа | Normoxia | Odds Ratio | P value |
|---------------------|---------|----------|------------|---------|
| | | | (95% CI) | |
| Primary Outcome | | | | |
| 30 day mortality | | | | |
| Secondary outcomes: | | | | |
| Adm. ICU 30 d | | | | |
| Reop. 30 d | | | | |
| Readm. 30 d | | | | |
| Blood 30 d | | | | |
| CRP | | | | |
| Creatinine | | | | |
| Troponine | | | | |

In order to assess the feasibility of the exposure groups, a supplementary sensitivity analysis will be made, reassessing the effect on outcome parameters when patients are reassigned to groups according to exposure to hypoxia  $\geq 8$  hours or hyperoxia  $\geq 8$  hours.

# OTHER INFORMATION

# **FUNDING**

This project has been funded by the internal grand for research projects at Bispebjerg and Frederiksberg Hospitals.

# APPENDIX 1



- 1. Hafner C, Wu J, Soto-Gonzalez L, et al. Moderate hyperoxia induces inflammation, apoptosis and necrosis in human umbilical vein endothelial cells. *Eur J Anaesthesiol*. 2017;34(3):141-149. doi:10.1097/EJA.000000000000593
- 2. Messina EJ, Sun D, Koller A, Wolin MS, Kaley G. Increases in oxygen tension evoke arteriolar constriction by inhibiting endothelial prostaglandin synthesis. *Microvasc Res*. 1994;48(2):151-160. doi:10.1006/mvre.1994.1046
- 3. Fonnes S, Gögenur I, Søndergaard ES, et al. Perioperative hyperoxia Long-term impact on cardiovascular complications after abdominal surgery, a post hoc analysis of the PROXI trial. *Int J Cardiol*. 2016;215:238-243. doi:10.1016/j.ijcard.2016.04.104
- 4. Meyhoff CS, Jorgensen LN, Wetterslev J, Christensen KB, Rasmussen LS. Increased long-term mortality after a high perioperative inspiratory oxygen fraction during abdominal surgery: Follow-up of a randomized clinical trial. *Anesth Analg*. 2012;115(4):849-854. doi:10.1213/ANE.0b013e3182652a51
- 5. Stub D, Smith K, Bernard S, et al. Air versus oxygen in ST-segment-elevation myocardial infarction. *Circulation*. 2015;131(24):2143-2150. doi:10.1161/CIRCULATIONAHA.114.014494
- 6. Cabello J, Burls A, Emparanaza J, Bayliss S, Quinn T. Oxygen therapy for acute myocardial infarction ( Review ). 2016;(12):49. doi:10.1002/14651858.CD007160.pub4.www.cochranelibrary.com
- 7. Manuel Wenk, MD, PhD, Hugo Van Aken, MD, PhD, and Alexander Zarbock, MD P. Oxygen friend or foe? *Anesth Analg.* 2017:Aug;125(2):682-687.
- 8. Pedersen NE, Rasmussen LS, Petersen JA, Gerds TA, Østergaard D, Lippert A. A critical assessment of early warning score records in 168,000 patients. *J Clin Monit Comput*. 2018;32(1):109-116. doi:10.1007/s10877-017-0003-5
- 9. Rasmussen JN, Rasmussen S, Gislason GH, et al. Mortality after acute myocardial infarction according to income and education. *J Epidemiol Community Health*. 2006;60(4):351-356. doi:10.1136/jech.200X.040972
- 10. Søgaard M, Madsen M, Løkke A, Hilberg O, Sørensen HT, Thomsen RW. Incidence and outcomes of patients hospitalized with COPD exacerbation with and without pneumonia. *Int J Chron Obstruct Pulmon Dis.* 2016:455. doi:10.2147/COPD.S96179
- 11. Kristensen PK, Thillemann TM, Pedersen AB, Søballe K, Johnsen SP. Socioeconomic inequality in clinical outcome among hip fracture patients: a nationwide cohort study. *Osteoporos Int*. 2017;28(4):1233-1243. doi:10.1007/s00198-016-3853-7
- 12. Meyhoff CS, Wetterslev J, Jorgensen LN, et al. Effect of High Perioperative Oxygen Fraction on Surgical Site Infection and Pulmonary Complications After Abdominal Surgery. *JAMA*. 2009;302(14):1543. doi:10.1001/jama.2009.1452
- 13. Ashby D. Practical statistics for medical research. Douglas G. Altman, Chapman and Hall, London, 1991. No. of pages: 611. Price: £32.00. *Stat Med*. 1991;10(10):1635-1636. doi:10.1002/sim.4780101015